CLINICAL TRIAL: NCT03329014
Title: A Randomized, Double-blind, Placebo-controlled 9-period Crossover, Dose-Escalation Study on the Safety, Bioavailability and Pharmacodynamics of Remimazolam Administered Intranasally as Powder and as Solution in Healthy Subjects
Brief Title: A Trial of Intranasal Remimazolam Pharmacokinetics, Pharmacodynamics, Safety and Bioavailability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paion UK Ltd. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNS7056-019
Record Dates: First submitted 2017-10-02; First posted 2017-11-01 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Procedural Sedation
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Intravenous Remimazolam (Experimental): 4 mg intravenous remimazolam as an intravenous control
  Interventions: Drug: Remimazolam
- 10 mg Powder Remimazolam (Experimental): Powder containing 10 mg remimazolam for intranasal administration
  Interventions: Drug: Remimazolam
- 10 mg Solution Remimazolam (Experimental): Solution containing 10 mg remimazolam for intranasal administration
  Interventions: Drug: Remimazolam
- 20 mg Powder Remimazolam (Experimental): Powder containing 20 mg remimazolam for intranasal administration
  Interventions: Drug: Remimazolam
- 20 mg solution Remimazolam (Experimental): Solution containing 20 mg remimazolam for intranasal administration
  Interventions: Drug: Remimazolam
- 40 mg Powder Remimazolam (Experimental): Powder containing 40 mg remimazolam for intranasal administration
  Interventions: Drug: Remimazolam
- 40 mg Solution Remimazolam (Experimental): Solution containing 40 mg remimazolam for intranasal administration
  Interventions: Drug: Remimazolam
- Placebo Powder (Placebo Comparator): Powder containing 20 mg placebo for intranasal administration
  Interventions: Drug: Placebo
- Placebo solution (Placebo Comparator): Solution containing 20 mg placebo for intranasal administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Remimazolam — For induction and maintenance of sedation
  Other Names: CNS7056
  Arms: 10 mg Powder Remimazolam; 10 mg Solution Remimazolam; 20 mg Powder Remimazolam; 20 mg solution Remimazolam; 40 mg Powder Remimazolam; 40 mg Solution Remimazolam; Intravenous Remimazolam
Drug: Placebo — Control arm
  Arms: Placebo Powder; Placebo solution

SUMMARY:
A prospective dose escalation, nine period cross-over trial assessing the safety, pharmacokinetics, bioavailability and pharmacodynamics of escalating doses of Remimazolam when administered intranasally as powder and solution in healthy subjects and compared to an intravenous control

DETAILED DESCRIPTION:
The design will be a randomized, double-blind, comparative, placebo- and active-controlled nine-period crossover study in healthy male volunteers. Subjects will be randomized and will receive each of the 9 treatments which will be separated by a minimum of 48 hours.The first treatment arm will always be the intravenous remimazolam. Eligible subjects will then be randomized to treatment sequence prior to study drug administration in treatment period 2. Each subject will participate in the study for up to 51 days, from Screening until Follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the trial, give written informed consent prior to the initiation of any protocol specific procedures, and to comply with the study restrictions.
2. Able to speak, read and understand English sufficiently to allow completion of all study assessments.
3. Gender: males
4. Age: 18 45 years, inclusive, at screening
5. Weight: 50 to 120 kg, inclusive, at screening
6. Body mass index: 19.0 to 33.0 kg/m2, inclusive, at screening
7. Healthy status, defined by the absence of evidence of any clinically significant, active or chronic diseases, in the opinion of the Investigator, following a detailed medical and surgical history, a complete physical examination, and evaluation of vital signs, 12 lead ECG, hematology, blood chemistry, serology, and urinalysis.
8. Previous experience with intranasal drug application (within the last year)
9. Ability and willingness to abstain from alcohol, caffeine, and xanthine containing beverages or food (e.g., coffee, tea, cola, chocolate, energy drinks) from 24 hours (1 day) prior to admission to the clinical facility on Day 0 until study discharge.
10. All values for hematology and for clinical chemistry tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the Investigator.

Exclusion Criteria:

1. Use of any intranasally applied medication within two weeks from randomization.
2. Use of benzodiazepines or other central nervous system (CNS) active drugs within 4 weeks of inclusion.
3. History of alcohol abuse or drug addiction (except nicotine), as defined by the Diagnostic and Statistical Manual of Mental Disorders, fifth edition, text revision (DSM V TR), or any self reported dependence or "addiction" within the subject's lifetime (except nicotine or caffeine).
4. Abnormal 12 lead ECG at screening, including:

   1. QTcF ≥ 450 ms
   2. QRS ≥ 110 ms
   3. PR ≥ 220 ms
   4. Second or third degree AV block
5. Use of any investigational drug or device within 30 days of the first dose of study medication.
6. History of relevant food allergies.
7. Any disease which, in the opinion of the Investigator, poses an unacceptable risk to the subjects.
8. Known allergy, hypersensitivity or prior intolerance to benzodiazepine derivatives or flumazenil, or a medical condition such that these agents are contraindicated.
9. Strenuous activity, sunbathing, and contact sports within 48 hours (2 days) prior to (first) admission to the clinical facility and for the duration of the study.
10. History of donation or loss of more than 450 mL of blood or blood products within 60 days prior to dosing in the clinical research center or planned donation before 30 days has elapsed since intake of study drug in the current study.
11. Positive screening test for hepatitis B surface antigen (HBsAg), anti hepatitis C virus (HCV) antibodies, or anti human immunodeficiency virus (HIV) 1 and 2 antibodies.
12. Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], barbiturates, benzodiazepines, tricyclic antidepressants and alcohol) at screening and at admission to the clinical research center; subjects positive for cannabinoids will be allowed only at the discretion of the Investigator.
13. Inability to be venipunctured or tolerate venous access as determined by the Investigator.
14. History of clinically significant, non remote suicidal ideations or suicide attempts based on the C SSRS that, in the opinion of the Investigator, pose an unacceptable risk to the subject for participating in the study.
15. Had had any major surgery within 4 weeks of study drug administration.
16. Requires concomitant treatment with any prescription or non prescription medications (with the exception of acetaminophen) or natural health products (herbal remedies), or respiratory depressants, or cannot safely discontinue these medications at least 7 days prior to receiving study drug.
17. Subject is an employee of the sponsor or research site personnel directly affiliated with this study or their immediate family member defined as a spouse, parent, child or sibling, whether biological or legally adopted.
18. A subject who, in the opinion of the investigator, is considered unsuitable or unlikely to comply with the study protocol for any reason.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-related Adverse Events | Predose until 180 minutes postdose
  Adverse events assessment will include: change in clinical laboratory assessments from baseline, change in vital signs from baseline, change in 12-lead electrocardiograms from baseline, drop in oxygen saturation measured using continuous pulse oximetry, nasal effect using the Nasal Effect Questionnaire (NEQ) and nose and throat examination. Adverse events with a respiratory or cardiovascular focus and adverse events related to effects seen with medications known to be associated with abuse will be analysed separately. The intensity, causality, outcome, seriousness and expectedness of adverse events will be assessed

SECONDARY OUTCOMES:
Alertness/Drowsiness using a bipolar 100-point Visual Analogue Scale (VAS) | Predose until 180 minutes postdose
  maximum effect (Emax), time to Emax (TEmax), minimum effect (Emin) and area under the effect curve (AUEC) determined pre-dose, 5, 10, 30, 60 and 180 minutes post dose
Agitation/Relaxation using a bipolar 100-point Visual Analogue Scale (VAS) | Predose until 180 minutes postdose
  maximum effect (Emax), time to Emax (TEmax), minimum effect (Emin) and area under the effect curve (AUEC) determined pre-dose, 5, 10, 30, 60 and 180 minutes post dose
Any Drug Effects using a unipolar 100-point Visual Analogue Scale (VAS) | Predose until 180 minutes postdose
  maximum effect (Emax), time to Emax (TEmax), minimum effect (Emin) and area under the effect curve (AUEC) determined pre-dose, 5, 10, 30, 60 and 180 minutes post dose
Memory/Amnestic Effects using the Paired Associates Learning (PALs) test | Predose until 180 minutes postdose
  maximum effect (Emax), time to Emax (TEmax), minimum effect (Emin) and area under the effect curve (AUEC) determined pre-dose,10, 30, 60 and 180 minutes post dose
Reaction Time using the Reaction Time Test | Predose until 180 minutes postdose
  maximum effect (Emax), time to Emax (TEmax), minimum effect (Emin) and area under the effect curve (AUEC) determined pre-dose, 20, 30, 60, 90, 120, 150 and 180 post dose
Time to Maximum Observed Plasma Concentration (Tmax) | From first dose of study drug until 240 minutes postdose
Maximum Observed Plasma Concentration (Cmax) | From first dose of study drug until 240 minutes postdose
Area Under the Plasma Concentration-time Curve from Zero to the last Measurable Concentration (AUC0-last) | From first dose of study drug until 240 minutes postdose
Area Under the Plasma Concentration-time Curve from Zero to Infinity (AUC0-∞) | From first dose of study drug until 240 minutes postdose
Terminal Elimination Half-life (t1/2) for Remimazolam and its Metabolite (CNS7054) | From first dose of study drug until 240 minutes postdose
Concentration at Time Zero (C0) for Intravenous Remimazolam and its Metabolite (CNS7054) Only | From first dose of study drug until 240 minutes postdose
The Fraction in Percent as a Measurement of the Rate and Extent to Which a Drug Reaches the Site of Action (F%) | From first dose of study drug until 240 minutes postdose
  F% will be calculated for the highest dose level (40 mg) and dose-proportionality will be evaluated across the dose range of 10 - 40 mg for each formulation (powder and solution) as available. Dose proportionality is AUC0-∞ and Cmax based. Bioavailability will be dose adjusted.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Searly, M.D, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No